CLINICAL TRIAL: NCT00948376
Title: Clinical and Molecular Study, Natural History of Asphyxiating Thoracic Dystrophy (DTJ)
Brief Title: Natural History of Asphyxiating Thoracic Dystrophy (DTJ)
Acronym: DTJ
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P060223
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-06

CONDITIONS: Asphyxiating Thoracic Dystrophy
Keywords: Natural history; IFT80; short ribs; multivisceral involvement
MeSH Terms: conditions — Jeune syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — phenotype-genotype
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: All ages
  Interventions: Genetic: IFT80 screening
- Fetuses
  Interventions: Genetic: IFT80 screening

INTERVENTIONS:
Genetic: IFT80 screening — Natural History
  Other Names: Natural History

SUMMARY:
The aim of the project is to prospectively analyze at a clinical and molecular level a series of 50 asphyxiating thoracic dysplasia (ATD) patients and 20 fetuses to further define the natural history of the disorder and to contribute to the identification of its molecular basis.

DETAILED DESCRIPTION:
Asphyxiating thoracic dysplasia (ATD, MIM 208500) belongs to the short rib polydactyly group and is characterized by short ribs often responsible for an early death due to respiratory distress, trident acetabular roof and short long bones.

In the course of the disease, renal, liver and eye complications may occur. However, their frequencies are unknown.

ATD is transmitted with an autosomal mode of inheritance and up till now only one gene has been identified, namely IFT80, which accounts only for a small part of ATD.

The aim of our project is to prospectively analyze at a clinical and molecular level a series of 50 ATD patients and 20 fetuses to further define the natural history of the disorder and to contribute to the identification of its molecular basis.

ELIGIBILITY:
Inclusion Criteria:

* Short ribs with narrow thorax
* Trident acetabular roof
* Short hands
* All ages
* Informed consent signed

Exclusion Criteria:

* Other disease
* Ellis van creveld syndrome
* No social security

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with:
  * Short ribs with narrow thorax
  * Trident acetabular roof
  * Short hands
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Natural history of asphyxiating thoracic dystrophy (ATD) | 3 years

SECONDARY OUTCOMES:
Correlation Phenotype-Genotype | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Cormier-Daire, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker, Paris, France